CLINICAL TRIAL: NCT05440890
Title: Early Treatment Based Neuroscience Education in Anterior Cruciate Ligament Repair Patients
Brief Title: Early Treatment Based Neuroscience Education in Knee
Acronym: ETbNE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Director, Clinical Research, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMAESHPhD
Record Dates: First submitted 2022-06-21; First posted 2022-07-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-06

CONDITIONS: Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Injuries
Keywords: cross-education; physiotherapy; unilateral strength training; fMRI; anterior cruciate ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, with two parallel groups (control and intervention)
Who Masked: Outcomes Assessor
Masking Description: Assessors are not aware of the allocation group of the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard protocol rehabilitation programme for an anterior cruciate ligament repair based on VAN MELICK N, et al 2016.
  Interventions: Other: Best current rehabilitation protocol
- Cross-education group (Experimental): Standard protocol rehabilitation programme for an anterior cruciate ligament repair based on VAN MELICK N, et al 2016.
  Additionally a contralateral lower limb strength training.
  Interventions: Other: Best current rehabilitation protocol; Other: Cross-training protocol

INTERVENTIONS:
Other: Best current rehabilitation protocol — Inflamation control and edema with physical agents, recover full pasive and active range of motion, normalize gait pattern, lower limb strengthening (specially quadriceps and hamstrings), neuromuscular control training, cycling, landings and running.
Other: Cross-training protocol — Beginning on 2º week after ACLR, 3 times per week during 8 weeks, based on isotonic exercise at least to 80% of 1RM in leg extension. 5 sets o 6 repetions with 1,5 - 2 minutes between series.
  Arms: Cross-education group

SUMMARY:
Determine the effecttiveness of a cross-education strength training protocol in a group of subjects with an anterior cruciate ligament surgery.

DETAILED DESCRIPTION:
The cross-education (CE) phenomenon has been studied in recent years as a form of gain muscle strength not only in healthy subjects but also in acute injuries such as musculoskeletal disorders and immovilitations. Unilateral training of the not injured limb has been suggested as an option to produce cross-edutation in terms of strength and skills. In addition, functional magnetic resonance imaging have been postulated as a promising tool to study the mechanisms of transfer.

In the context of our study, arthrogenic muscle inhibition (AMI) of knee extensors is a common consequence after ACL repair in which a CE strength training can lead to reduce quadriceps atrophy and its implications in long terms achievements. Thus, an unilateral strength protocol of the uninjuried limb, according to the last Delphi Consensus, will be run for 8 weeks to check the possible benefits of the transfer in a sample of ACL repair.

ELIGIBILITY:
Inclusion Criteria:

* People between 18 and 40 years whith MRI diagnosis of ACL rupture.
* Autograft, allograft or artificail graft of any source.
* With/without any meniscal resection/repair.

Exclusion Criteria:

* Diagnosis of systematic disease, no injury or symptomatic in contralateral lower limb, pregnancy, current or prior neurologic condiction.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Changes in quadriceps strength. | Baseline and 12 weeks post-surgery
  Isometric Maximal voluntary contraction in 60º/90º of knee flexion. Both legs. Patients performed two familiarization trials at 50% of their estimated MVC. Then 3 test of maximal contraction will be done. Measured in newtons.
Changes in cortical adaptation. | Baseline and 10 weeks post-surgery
  Functional magnetic resonance including tractography, blood oxygen level dependent (BOLD) and resting-state study to measure how and where the cortical activation is meanwhile the subjects perform a 50% of the MVIC of knee extension with the injuried leg. Special focus on primery motor cortex and supplementary motor area.

SECONDARY OUTCOMES:
Limb symmetry index (LSI). | Pre- surgery, 12 weeks post-surgery
  Comparison of both quadriceps MVC. Measured in percentage.
Peak rate of force development (RFD). | Pre- surgery, 12 weeks post-surgery
  Explosive strength as the speed which the muscle (quadriceps) can develop force. Measured in newtons per second.
Muscle activation. | Pre- surgery, 12 weeks post-surgery
  Surface eletromyography in the main muscles of lower limb (rectus femoris, vastus medialis, vasto lateralis, biceps femoris) during the MVC test and functional task such as active straigth leg raise, gait, bilateral/unilateral squat, bilateral/unilateral rumanian deadlift, lunges and single and normal countermovement jump.
Cross-sectional area of quadriceps | Pre- surgery, 12 weeks post-surgery
  Sonography of quadriceps to determine the cross-sectional area of rectus femoris, vastus medialis and vastus laterlis. Measured in cm2.
The International Knee Documentation Committee (IKDC) questionnarie. | 12 weeks post-surgery
  IKDC is a reliable and valid measure for ACLR. It consists on 10 items related to knee symptons, knee function and sports activities. Score range from 0 to 100 with higher scores determine less disfunction.
The Lysholm questionnaire. | 12 weeks post-surgery
  Total score of 100 points including the following variables: crutch support, knee locking, knee instability, pain, swelling and knee function. Score range 0 to 100 with high scores indicating better and positive knee outcomes.
The Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire. | 12 weeks post-surgery
  The KOOS is a self-administered questionnaire with variables related to symptons, pain, quality of life, daily tasks and function and sport activities. Score range 0 to 100 with high scores indicating better and positive knee outcomes.
Muscle thickness of quadriceps. | Pre- surgery, 12 weeks post-surgery
  Measured in cm by ultrasonography in both quadriceps.
Step length during gait | 12 weeks post-surgery
  Measured in cm of each limb with Optogait system.
Contact time with the ground during gait | 12 weeks post-surgery
  Measured in seconds of each limb with Optogait system
Cadence of the gait | 12 weeks post-surgery
  Measured in step per seconds with Optogait system

REFERENCES:
- [Background] Manca A, Hortobagyi T, Carroll TJ, Enoka RM, Farthing JP, Gandevia SC, Kidgell DJ, Taylor JL, Deriu F. Contralateral Effects of Unilateral Strength and Skill Training: Modified Delphi Consensus to Establish Key Aspects of Cross-Education. Sports Med. 2021 Jan;51(1):11-20. doi: 10.1007/s40279-020-01377-7. PMID 33175329
- [Result] Cuyul-Vasquez I, Alvarez E, Riquelme A, Zimmermann R, Araya-Quintanilla F. Effectiveness of Unilateral Training of the Uninjured Limb on Muscle Strength and Knee Function of Patients With Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-Analysis of Cross-Education. J Sport Rehabil. 2022 Mar 12;31(5):605-616. doi: 10.1123/jsr.2021-0204. Print 2022 Jul 1. PMID 35279020